CLINICAL TRIAL: NCT02748122
Title: A Clinical Pilot to Assess Feasibility of Using Continuous Subcutaneous Insulin Injection Therapy (CSII: Insulin Pump) in Adolescents With Type 2 Diabetes (T2DM)
Brief Title: CSII Pilot in Adolescents With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00313
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetes
Keywords: Adolescents; Insulin; T2DM
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with T2DM (Experimental)
  Interventions: Other: MMT 723

INTERVENTIONS:
Other: MMT 723 — Subjects will have the insulin pump inserted. With the aid of a small needle, the catheter (tube) of the insulin pump will be inserted through the skin into fatty tissue and will be taped in place. The subject will be required to wear the pump for three (3) months.

SUMMARY:
This feasibility pilot is intended to understand whether adolescents with Type 2 Diabetes (2DM) can be transitioned to a continuous subcutaneous insulin injection (CSII) and if so, assess whether CSII is a feasible treatment modality and improves quality of life (QOL) in adolescents with T2DM over 3 month period.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with Type 2 Diabetes mellitus between the ages of 12- 23 years, who have had T2DM for at least 6 month duration, and who have had a HbA1c > 8% in the preceding 3 months prior to enrollment into the study. As a diabetes is a chronic disease the AAP (American Academy of Pediatrics; 2002) definition of a "Pediatric patient "is from birth until 21 years old. There are patients in the Diabetes program that we sometimes follow for 2-3 years beyond this age of 21 years and therefore would like to offer this study until the age of 23 years. This will give opportunity to our patients to be recruited if they would choose to participate in the study.
* Confirmed T2DM as defined by American Diabetes Association i.e. FPG > 126 mg/dL or blood sugar > 200 mg/dl on a 2 hr, 75 g OGTT or random blood sugar >200 mg/dl. Pubertal, Tanner stage >1
* Subjects must be willing to comply with study protocol requirements
* Females must have a negative pregnancy test within 72 hours prior to the start of the study and on every subsequent study visit. If on any visit their pregnancy test is positive they will be asked to not continue in the study. If the adolescent is using contraception such as birth control pills they will be allowed to continue using them during the study as this should not affect glucose levels. Once a female is confirmed to be pregnant we will take the insulin pump and restart insulin injection regimen that they were before the start of the study. We will also make an aptt with "high risk obstretics" and encourage the adolescent to check their blood sugars at least 4-6 times per day.
* The patient must be on insulin to qualify for the study. The adolescents could be on oral hypoglycemic agent in addition to insulin to be included in the study.

Exclusion Criteria:

* Chart review of adolescents with T2DM will be done to confirm absence of glutamic acid decarboxylase, islet cell or insulin autoantibodies or secondary causes of diabetes
* Other significant major organ system illness
* Females who are pregnant at their initial assessment. We will be testing female participants on every visit with a urine pregnancy test and if they are found to pregnant we will ask them to stop using their pump and go back to using insulin injections.
* Significant psychiatric illness: schizophrenia, bipolar disorder, active substance abuse and uncontrolled major depression.
* All adolescents who have signs of renal insufficiency (creatinine clearance based on Schwartz equation >0.55 for females and males 0.7 ages 13-18 years) (13). Serum creatinine will be available on the metabolic profile. Subjects with elevated CrCl will be excluded from the study.

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Change in score on Quality of Life questionnaire | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Preneet Brar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States